CLINICAL TRIAL: NCT06671587
Title: A 20-week, Multicenter, Prospective, Parallel-group Treatment, Open-label, 2-Arm, Phase 4, Randomized Study to Evaluate the Efficacy of iGlarLixi Versus Gla-100 on Glycemic Time in Range (TIR) From Continuous Glucose Monitoring (CGM) in Chinese Insulin Naïve Patients With Type 2 Diabetes (T2D) Inadequately Controlled With Oral Antidiabetics
Brief Title: iGlarLixi CGM Study in Chinese T2D Individuals After OADs
Acronym: China Soli-CGM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS18034; U1111-1306-6660 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes (T2D)
Keywords: Glucagon-like peptide-1 receptor agonist (GLP-1 RA); FRC (fixed ration combination)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide

STUDY DESIGN:
Intervention Model Description: Open-label, 1:1 randomized, active-controlled, 2-arm, 20-week treatment duration, parallel-group, multicenter, phase IV study comparing iGlarLixi to Gla-100.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iGlarLixi (insulin glargine/lixisenatide) (Experimental): Participants will receive iGlarLixi once daily for 20 weeks. iGlarLixi is to be initiated with the starting daily dose of 5-10 dose steps on Visit 4 (Day 1) and will be titrated according to fasting SMBG to achieve glycemic target of ≥80 and ≤110 mg/dL.
  Interventions: Drug: iGlarLixi (insulin glargine/lixisenatide)
- Gla-100 (insulin glargine) (Active Comparator): Participants will receive Gla-100 once daily for 20 weeks. Gla-100 is to be initiated with the starting daily dose of 5-10 U on Visit 4 (Day 1) and will be titrated according to fasting SMBG to achieve and maintain same glycemic target of ≥80 and ≤110 mg/dL.
  Interventions: Drug: Gla-100 (insulin glargine)

INTERVENTIONS:
Drug: iGlarLixi (insulin glargine/lixisenatide) — iGlarLixi will be supplied as a sterile aqueous solution in a pen-injector.
  There will be 2 pen-injectors with different insulin glargine/lixisenatide fixed ratios which allow insulin glargine titration from 5 U/day to 40 U/day while limiting lixisenatide dose to a maximum of 20 μg/day:
  - iGlarLixi must not be mixed with other insulins nor diluted.
  Other Names: SOLIQUA®
  Arms: iGlarLixi (insulin glargine/lixisenatide)
Drug: Gla-100 (insulin glargine) — Gla-100 will be supplied as a 3 mL sterile aqueous solution for SC injection in a pre-filled disposable Gla-100 SoloStar® pen containing 300 U insulin glargine (100 U/mL). Doses could be set in the range of 5 to 80 U in increments of 1 unit.
  Other Names: LANTUS®
  Arms: Gla-100 (insulin glargine)

SUMMARY:
This study is an open-label, 1:1 randomized, active-controlled, 2-arm, 20-week treatment duration, parallel-group, multicenter, phase IV study to evaluate the effect of iGlarLixi versus Gla-100 on glycemic control measured as TIR from CGM device in Chinese insulin naïve patients with T2D inadequately controlled with OADs. At the end of the screening period, eligible participants will be randomized to one of two treatment groups (iGlarLixi or Gla-100 group). The randomization (1:1) will be stratified by values of HbA1c at screening (<8.0%, ≥8.0%), and background treatment (metformin only, metformin+SGLT-2i).

Study details include:

* The study duration per participant will be approximately up to 24 weeks.
* The treatment duration will be up to 20 weeks.
* The number of visits will be 14 visits including 9 times of on-site visits and 5 times of phone call visits in total during screening and treatment periods. On-site every 1 week will be from screening till randomization (Week 0), then on site or phone call visit every 2 weeks till Week 12, then every 3 weeks till Week 18, and the End of Treatment visit will be conducted at Week 20. There will be a safety follow-up by a phone call visit (End of Study) in 3 days (-1/+3 days) after the last dose of the treatment.
* Health measurement/Observation: change in TIR as the primary endpoint
* Intervention name: iGlarLixi and Gla-100
* Participant gender: male and female
* Participant age range: adults at least 18 years of age
* Condition/disease: type 2 diabetes
* Study hypothesis: compared to Gla-100, iGlarLixi will demonstrate a superiority therapeutic effect on glycemic control assessed by change in TIR measured with CGM from baseline to Week 20 in the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed as T2D of at least 1 year before screening visit
* Participants who are treated at least 3 months prior to screening visit with a stable dose of metformin alone or in combination with a second OAD
* Inadequate control
* Body mass index (BMI) within the range 20-40 kg/m2 (inclusive)
* Is willing and able to wear the CGM device continuously
* Is willing to discontinue daily (oral) SU, glinide, alpha-GI, and DPP-4i
* Not using another CGM device during the study

Exclusion Criteria:

* Participants with severe renal dysfunction
* Participants with short life expectancy
* Participants with conditions/concomitant diseases making them non evaluable for the efficacy endpoints
* Participants with conditions/concomitant diseases precluding their safe participation in this study
* An episode of severe hypoglycemia requiring the assistance of a third party within 3 months before screening visit
* History of clinically significant pancreatitis or severe gastrointestinal disorders
* Participants who have any history of severe multiple allergies or an allergy resulting in anaphylaxis, or contraindication/hypersensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study
* Previous treatment with insulin
* Use of any glucose-lowering agents other than metformin alone or in combination with a second OAD (can be a SU, a glinide, an alpha-GI, a DPP-4i, or a SGLT-2i)
* Use of systemic glucocorticoids
* Use of weight loss drugs
* History of discontinuation of a previous treatment with GLP-1 RA for safety/tolerability reasons or lack of efficacy
* Laboratory findings at the screening visit
* Participants have any current or previous skin conditions
* Participants unwilling or unable to do blood glucose monitoring using the Sponsor-provided blood glucometer at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Superiority of mean change in the percentage of TIR [3.9-10.0 mmol/L (70-180 mg/dL)] | from baseline to Week 20
  Superiority of mean change in the percentage of TIR [3.9-10.0 mmol/L (70-180 mg/dL)] from baseline to Week 20 of iGlarLixi vs Gla-100

SECONDARY OUTCOMES:
2a Proportion (%) of participants achieving TIR target as >70% | Week 20
2b Change (%) in TAR >10.0 mmol/L (>180 mg/dL) | from baseline to Week 20
2c Change (mg/dL) in mean daily glucose | from baseline to Week 20
2d Proportion (%) of participants achieving composite target of TIR as >70% [3.9-10.0 mmol/L (70-180 mg/dL)] with TAR as <25% [>10.0 mmol/L (>180 mg/dL)] with TBR as <4% [<3.9 mmol/L (<70 m)/dL)] | Week 20
Change (%) in coefficient of variation (CV) | from baseline to Week 20
Change (%) in the percentage of time in tight range (TITR) [3.9-7.8 mmol/L (70-140 mg/dL)] | from baseline to Week 20
Proportion (%) of participants achieving TITR [3.9-7.8 mmol/L (70-140 mg/dL)] >50% | Week 20
Proportion (%) of participants achieving ≥5% TIR improvement | from baseline to Week 20
Proportion (%) of participants achieving ≥10% TIR improvement | from baseline to Week 20
Change (%) in TAR >13.9 mmol/L (>250 mg/dL) | from baseline to Week 20
Change (%) in time below range (TBR) | from baseline to Week 20
  * <3.9 mmol/L (<70 mg/dL), including <3.0 mmol/L (<54 mg/dL)
  * <3.0 mmol/L (<54 mg/dL)
  * <3.9 mmol/L (<70 mg/dL), including <3.0 mmol/L (<54 mg/dL) in nocturnal (00:00 h-05:59 h) time
  * <3.0 mmol/L (<54 mg/dL) in nocturnal (00:00 h-05:59 h) time
Change in mean glucose standard deviation (SD) | from baseline to Week 20
Change (%) in glucose management indicator (GMI) | from baseline to Week 20
Proportion (%) of participants achieving CV <36% | Week 20
Proportion (%) of participants achieving CV <32% | Week 20
Change (%) in HbA1c | from baseline to Week 12 and Week 20
Proportion (%) of participants achieving HbA1c <7% | Week 12 and Week 20
Proportion (%) of participants achieving HbA1c <7% without documented hypoglycemia | Week 20
  documented hypoglycemia (defined as ADA Level 1, 2 or 3)
Proportion (%) of participants achieving HbA1c <7% without body weight gain | Week 20
  body weight gain (≥5% compared to baseline)
Proportion (%) of participants achieving HbA1c <7% without documented hypoglycemia and without body weight gain | Week 20
  documented hypoglycemia (defined as ADA Level 1, 2 or 3)
Change (mmol/L) in fasting plasma glucose (FPG), 2-hour postprandial glucose (PPG) | from baseline to Week 12 and Week 20
Change (nmol/L) in fasting C-peptide and post-prandial C-peptide | from baseline to Week 12 and Week 20
Change (U and U/Kg) in insulin dose | from baseline to Week 20
Change (kg) in body weight | from baseline to Week 20
Change (%) in TIR [3.9-10.0 mmol/L (70-180 mg/dL)], TAR [>10.0 mmol/L (>180 mg/dL)] and TBR [3.0 mmol/L (<54 mg/dL)] for specific time blocks (6 am-12 pm, 12 pm-6 pm, 6 pm-12 am, and 12 am-6 am) | from baseline to Week 20
Change in diabetes medication treatment satisfaction scores (total score and by subscales), using the treatment-related impact measure diabetes (TRIM-D) questionnaire | from baseline to Week 20
AE, serious adverse event (SAE), and adverse event of special interest (AESI) | from screening to week 21
Overall hypoglycemia events and rates | from screening to week 21
Nocturnal (00:00 h-05:59 h) hypoglycemia events and rates | from baseline to Week 20
Confirmed hypoglycemia (ADA Level 1, 2 and 3) | from baseline to Week 20
  * ADA Level 1: Measurable glucose concentration <70 mg/dL (3.9 mmol/L) but ≥54 mg/dL (3.0 mmol/L)
  * ADA Level 2: Measurable glucose concentration <54 mg/dL (3.0 mmol/L) that needs immediate action
  * ADA Level 3: Severe event characterized by altered mental and/or physical functioning that requires assistance from another person for recovery

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number: 1560001, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org